CLINICAL TRIAL: NCT05633329
Title: Comparison Between the Efficacy of Ultrasound Guided Single Injection Erector Spinae Plane Block Versus Dual Injection Erector Spinae Plane Block for Postoperative Pain in Patients Undergoing Abdominal Surgery: Randomized Clinical Study
Brief Title: Dual Injection ESPB Versus Single Injection ESPB for Laparotomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hassan Mokhtar Elshorbagy Hetta, lecturer of anesthesia and ICU, Minia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 474:10/2022
Record Dates: First submitted 2022-11-04; First posted 2022-12-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain; Regional Block
Keywords: ESPB; pain; regional block
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Floors and Floorcoverings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single ESPB (Experimental): single injection at level T8
  Interventions: Procedure: single level
- dual ESB (Experimental): dual injection at level T7 and T9
  Interventions: Procedure: dual level

INTERVENTIONS:
Procedure: single level — injection of 40 ml bupivacaine 0.25 at T8 (20 ml on each side)
  Arms: single ESPB
Procedure: dual level — injection of 40 ml of bupivacaine 0.25 at two level T7 and T9 (10 ml on each level of both side)
  Arms: dual ESB

SUMMARY:
To evaluate and compare the efficacy of single level injection erector spinae plane block versus double level injection Erector spinae plane block in laparotomies

ELIGIBILITY:
Inclusion Criteria:

1. Age18-60.
2. Both genders.
3. abdominal surgery.
4. ASA I-III.

Exclusion Criteria:

1. Drug allergy.
2. Morbid obesity (BMI >40 kg/m2).
3. Psychiatric disorder.
4. Opiod dependence.
5. patient refuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
first analgesic request | 24 hours
  time to request fentanyl

SECONDARY OUTCOMES:
resting visual analogue pain scale | 24 hours
  pain score at rest from 0-10 which 0 mean no pain and 10 the worst pain
dynamic visual analogue pain scale | 24 hours
  pain score at movement (cough) from 0-10 which 0 mean no pain and 10 the worst pain
analgesic consumption | 24 hours
  total fentanyl required first day postoperative

CONTACTS AND LOCATIONS:
Overall Officials: hassan m. hetta, lecturer, Principal Investigator — Minia University, faculty of medicine
Locations (1):
- Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No